CLINICAL TRIAL: NCT01145989
Title: A Phase II Study of AT9283 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of AT9283 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I191
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — 1-cyclopropyl-3-(3-(5-morpholin-4-ylmethyl-1H-benzoimidazol-2-yl)-1H-pyrazol-4-yl)urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AT9283 (Experimental): Starting dose will be 40 mg/m2/day OR 30 mg/m2/day to be confirmed at registration. IV 24 hour continuous infusion Days 1 and 8 every three weeks
  Interventions: Drug: AT9283

INTERVENTIONS:
Drug: AT9283 — Starting dose will be 40 mg/m2/day OR 30 mg/m2/day to be confirmed at registration. IV 24 hour continuous infusion Days 1 and 8 every three weeks

SUMMARY:
The purpose of this study is to find out whether the new drug AT9283 will slow the growth of multiple myeloma. Side effects of AT9283 will also be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of multiple myeloma, according to the internationally accepted criteria for myeloma [International Myeloma Working Group 2003], must have been made prior to initial treatment.
* Patients must have measurable disease, according to the internationally accepted criteria for myeloma [Durie 2006].
* Age ≥ 18 years.
* ECOG performance status of 0, 1 or 2.
* Life expectancy > 3 months.
* Patients must have received prior treatment for multiple myeloma and have relapsed or progressed on prior therapy. There is no limit on number of prior treatment regimens, but patients must have completed prior treatment at least 4 weeks prior to registration (< 4 weeks permitted if prior therapy is non-myelosuppressive or if any treatment-related myelosuppression has resolved. Please call NCIC CTG for discussion). Patient must have recovered from any treatment related adverse events.
* In patients with significant cardiac history or prior anthracycline exposure, Left Ventricular Ejection Fraction (LVEF) must be ≥ 50%.
* Prior radiation is permitted, but must have been completed at least 4 weeks prior to registration. Exceptions may be made for low dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG.
* Laboratory Requirements: (must be within 7 days prior to registration) Hematology: Absolute granulocytes (AGC) ≥ 1.0 x 109/L Platelets ≥ 70 x 109/L Hemoglobin >100 g/L Biochemistry: Serum creatinine ≤ 1.5 x ULN Bilirubin normal AST and ALT ≤ 2 x upper normal limit Calcium normal
* In patients with significant cardiac history or prior anthrecycline exposure, left-ventricular ejection fraction (LVEF) must be ≥ 50%
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is provided. A copy of the initial REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to randomization or registration. Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial.
* Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, toxicity, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

* Patients with uncontrolled hypertension (resting BP consistently higher than systolic > 140 mmHg and/or diastolic > 90 mmHg)
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, prostate cancer with stable PSA for ≥ 3 years, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test within 7 days prior to registration and must be using effective contraception throughout the study.
* Patients receiving concurrent treatment with other anti-cancer therapy.
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit that patient to be managed according to the protocol.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects) are not eligible.
* Patients with uncontrolled hypertension (resting BP> 140 mmtlg and/or diastolic > 90 mmtlg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2015-11-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years

SECONDARY OUTCOMES:
Adverse effects of AT9283 | 3 years
Evaluation of potential predictive and prognostic biomarkers (marrow, blood) | 3 years
Evaluation of disease-related symptoms including pain, fatigue, mucositis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tony Reiman, Study Chair — Atlantic Health Sciences Corporation, Saint John Regional Hospital
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hay AE, Murugesan A, DiPasquale AM, Kouroukis T, Sandhu I, Kukreti V, Bahlis NJ, Lategan J, Reece DE, Lyons JF, Sederias J, Xu H, Powers J, Seymour LK, Reiman T. A phase II study of AT9283, an aurora kinase inhibitor, in patients with relapsed or refractory multiple myeloma: NCIC clinical trials group IND.191. Leuk Lymphoma. 2016;57(6):1463-6. doi: 10.3109/10428194.2015.1091927. Epub 2015 Oct 15. No abstract available. PMID 26376958